CLINICAL TRIAL: NCT02045498
Title: Effect of Capnography Feedback During Cardiopulmonary Resuscitation on Quality Performance of Rescuers and Outcome of the Patient
Brief Title: Effect of Capnography Feedback During Cardiopulmonary Resuscitation (CPR ) on Patient's Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyedreza Mazloum, dr seyed reza mazlom, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: capnography feedback
Record Dates: First submitted 2014-01-19; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Cardiopulmonary Arrest
Keywords: cpr; feedback; capnography; outcome; quality; resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- capnography, feedback, quality of cpr (Experimental): capnography feedback was used for management of the resuscitation and quality of cpr performance in rescuers and outcomes of the patients was measured.
  Interventions: Device: capnography feedback
- conventional cpr (No Intervention): conventional cpr

INTERVENTIONS:
Device: capnography feedback — capnography feedback was used for management of the resuscitation and quality of cpr performance in rescuers and outcomes of the patients was measured.
  Arms: capnography, feedback, quality of cpr

SUMMARY:
Compare the quality performance of rescuers and resuscitation outcomes of cardiac arrest patients in both groups with and without capnography feedback

DETAILED DESCRIPTION:
This study has done at Mashhad Ghaem Educational center. Two nurses and an anesthesia resident selected and trained according to the latest guidelines of CPR . In the control sample, with the declare of code 99 and attend the team on the patient's bedside, CPR begins and then every two minutes, return of the patient checks in the usual way. quality performance of rescuers ,Recovery or death of the patient and the result is recording. In the second phase , group members were educated how to use capnography (Comdek's MD-660P Oxi-Capnography) in CPR and guiding restoration efforts by it. with the code 99 and attend the team on the patient's bedside capnography uses and its waveforms will appear on the monitor device which is visible to all rescuers and the quality of performance is renewed based on the its guidance. The two groups patients for age, sex, initial rhythm of arrest, time of arrest until the first action, the time of arrest until the first shocks are comparing to control these factors influence on the outcome. quality performance of rescuers , resuscitation outcomes and CPR duration and relative factors in each of the groups were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest patient age more than 18

Exclusion Criteria:

* age more than 80 cardiac arrest due to pulmonary embolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
chest compressions and artificial ventilation rate in a minute | By the end of twenty minutes of CPR
  The number Of chest compressions and artificial ventilation rate in a minute by rescuers in both study groups (with and without capnography feedback) were assessed.

SECONDARY OUTCOMES:
Return of spontaneous circulation or death of patient at the end of resuscitation | about twenty minutes After start of CPR
  Return of spontaneous circulation or death of patient at the end of resuscitation in both study groups (with and without capnography feedback) were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tayebe PourGhaznein, MSc, Study Director — MUMS
Locations (1):
- Ghaem Educational, Research and Treatment Center, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Background] Qvigstad E, Kramer-Johansen J, Tomte O, Skalhegg T, Sorensen O, Sunde K, Olasveengen TM. Clinical pilot study of different hand positions during manual chest compressions monitored with capnography. Resuscitation. 2013 Sep;84(9):1203-7. doi: 10.1016/j.resuscitation.2013.03.010. Epub 2013 Mar 15. PMID 23499897
- See also: In-hospital Cardiac Arrest: Catching up with Advances Made in Out-Of-Hospital Cardiac Arrest — http://www.heart.org/HEARTORG/